CLINICAL TRIAL: NCT01086371
Title: Rhythmic Auditory Stimulation and Walking Performance in MS Patients
Brief Title: Rhythmic Auditory Stimulation and Walking Performance in Multiple Sclerosis (MS) Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study being redesigned in anticipation of new study protocol.
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Francois Bethoux, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAS Gait MS
Record Dates: First submitted 2010-01-29; First posted 2010-03-15 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Gait Disturbance in Multiple Sclerosis Patients
Keywords: Multiple Sclerosis; gait
MeSH Terms: conditions — Multiple Sclerosis | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- RAS walking (Experimental): Subjects will walk while listening to music 20 minutes per day every day during the study period.
  Interventions: Other: Rhythmic auditory stimulation; Other: Walking exercise
- RAS no walking (Active Comparator): Subjects will be listening to music but not performing walking exercise, for 20 minutes per day every day during the study period.
  Interventions: Other: Rhythmic auditory stimulation
- Walking no RAS (Active Comparator): Subjects will be walking without listening to music for 20 minutes per day every day during the study period
  Interventions: Other: Walking exercise

INTERVENTIONS:
Other: Rhythmic auditory stimulation — Recorded music with embedded beat set 10% above the subject's baseline walking cadence.
  Other Names: Rythmic Auditory Stimulation, RAS, Music
  Arms: RAS no walking; RAS walking
Other: Walking exercise — Subjects will be walking daily for a total of 20 minutes (may be broken down to smaller time periods.
  Other Names: Walking
  Arms: RAS walking; Walking no RAS

SUMMARY:
The study is being conducted to determine if a home-based walking program that uses RAS (Rhythmic Auditory Stimulation)is a viable and effective treatment of gait instability for people with MS.We hypothesize that an RAS-based home walking program will demonstrate significant improvements over both regular exercise and no exercise. To test this hypothesis we will compare between group differences from baseline and three weeks of intervention on 3 quantitative gait measures and 1 standardized MS measurement from the following 3 groups: RAS walking, RAS no walking Other: Walking exercise The secondary goal of the study will be to determine any carry-over effects of RAS on gait parameters in ambulatory patients with MS. We hypothesize that RAS will produce sustained changes in gait pattern due to entrainment processes. To test this hypothesis, we will compare gait parameters two weeks following the cessation of the intervention with baseline and with the last week of intervention.

The third goal of this study is to determine if RAS-enhanced exercise has any transfer to improve other areas such as upper extremity function and/or cognitive function. We hypothesize that those participating in an RAS-based home walking program will demonstrate improvements in other domain areas, such as cognitive and upper body functioning. To test this hypothesis we will compare results from the Multiple Sclerosis Functional Composite(MSFC) taken at baseline and again at the end of the treatment phase for all three groups.

DETAILED DESCRIPTION:
Thirty three patients will be recruited for the study.There will be three study groups 1)the walking and music group,2)music only no walking group 3)walking only no music group The subjects in the walking + music group and the music - no walking group will be provided a list of songs to choose from. MP3 players will be provided that contain the chosen music, which has been altered electronically with an embedded beat and set to their baseline walking cadence +10%. The subjects in the walking + music group will be instructed to walk while listening to the music for 20 minutes per day every day. The subjects in the music - no walking group will be instructed to sit in a chair and listen to the music for 20 minutes per day every day. The subjects in the walking -no music group will be instructed to walk for 20 minutes per day every day. The total duration of the interventions will be 3 weeks.

Study schedule Visit 1 (baseline): informed consent will be obtained. Subjects will be screened for inclusion/exclusion criteria.Subjects qualified for the study will be randomized to the treatment (MT) or control (C) group. Baseline assessments will be performed on all subjects.Subjects in the walking+music group and the music- no walking group will be given mp3 players with music.

Visit 2 (week 3): assessments will be performed on all subjects.All subjects will be instructed to discontinue walking and music regimens.

Visit 3 (week 5): All subjects will return for final assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of multiple sclerosis documented in medical records
* Able to walk at least 100 feet without physical assistance (use of assistive devices such as cane, crutch, or walker is allowed.

Exclusion Criteria:

* Treatment for an MS exacerbation in the past 30 days
* Severe co morbidity precluding participation in the study per investigator's judgment (e.g. severe cardiac or respiratory failure)
* Severe cognitive deficits precluding informed consent or preventing the subject from following study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Stride Length | each study visit: baseline, week 3, and week 5 a total of 3 visits over a 5 week period of time

SECONDARY OUTCOMES:
25 foot walk time | each study visit: baseline, week 3, and week 5 a total of 3 visits over a 5 week period

CONTACTS AND LOCATIONS:
Overall Officials: Francois A Bethoux, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States